CLINICAL TRIAL: NCT06927843
Title: A Cross-sectional Investigational Study to Evaluate the Sensitivity, Specificity, and Utility of the DPP® Syphilis Screen & Confirm Antibody Point-of-care Test (POCT) to Diagnose Infectious Syphilis in Participants Attending the Nine Circles Community Health Centre in Winnipeg, Manitoba
Brief Title: Investigational Study to Evaluate the DPP® Syphilis Screen & Confirm Antibody Point-of-care Test (POCT) to Diagnose Infectious Syphilis
Status: Recruiting | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government); Chembio Diagnostic Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HS26266
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Syphilis
Keywords: syphilis; Point of Care Test; Serology
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: point of care test — DPP Syphilis Screen and Confirm antibody point-of-care-test (POCT)

SUMMARY:
The goal of this observational study is to evaluate the sensitivity, specificity, and utility of the DPP® Syphilis Screen & Confirm antibody point-of-care test (POCT) to diagnose infectious syphilis in participants attending the Nine Circles Community Health Centre in Winnipeg, Manitoba.

The main questions are: Does the POCT provide accurate results compared to conventional syphilis serology methods? and Can the use of POCT improve the timeline for diagnosis and treatment of syphilis?

Researchers will compare the POCT results with conventional laboratory testing to assess if the rapid test can reliably diagnose syphilis during the initial clinic visit.

Participants will: Provide a blood sample via fingerstick for POCT testing and complete a feedback survey to evaluate the POCT experience.

Key details: This study will involve approximately 600 participants aged 18 and older over the course of 12 months which includes both new and repeat visits

ELIGIBILITY:
Inclusion Criteria:

* Individuals attending the Clinic for routine sexual health care and requiring syphilis testing as part of this care
* Be able to provide informed consent and are a minimum 18 years of age are eligible for this study
* Those who had other STIs in the past, or being suspected of having other STIs, are not excluded as long as testing for syphilis is part of the care provided to them

Exclusion Criteria:

* Those who, at the discretion of the HCP/Research Nurse, appear intoxicated and/or with extreme distress, or confused, will be excluded
* Those below the age of 18 years
* if it has been less than 90 days since their last POCT study visit and they are asymptomatic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population for this research comprises individuals seeking care at the Nine Circles Community Health Centre in Winnipeg, Manitoba, Canada. Participants are adults (aged 18 years or older) attending the clinic for routine sexual health care, which includes syphilis testing as part of their standard care. The clinic caters to a diverse urban population which is comprised of newcomers to Canada, indigenous, and LGBTQ2S+ community and receives a significant number of syphilis serology specimens annually, reflecting a broad spectrum of individuals who may present with varying sexual health needs. This setting provides a unique opportunity to evaluate the performance of the DPP® Syphilis Screen & Confirm antibody point-of-care test in a real-world clinical environment
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Point of Care Test Performance | From start of enrollment to the end of the enrollment period (12 months)
  Sensitivity of POCT: Percentage of participants with laboratory-confirmed active syphilis who are identified as positive by the POCT, Specificity of POCT: Percentage of participants without laboratory-confirmed active syphilis who are identified as negative by the POCT

SECONDARY OUTCOMES:
Secondary POCT Performance Measures | From start of enrollment to the end of the enrollment period (12 months)
  False Positive Rate: Percentage of participants without active syphilis who test positive by POCT for active syphilis. False Negative Rate: Percentage of participants with active syphilis who test negative by POCT for active syphilis.
Comparison of Results by POCT Methodology | From start of enrollment to the end of the enrollment period (12 months)
  Comparison of visual vs micro-reader assisted results

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — University of Manitoba
Locations (1):
- Nine Circles Community Health Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Data and information will not be shared outside agencies for safety and privacy of the participants. Performance of POCT will be evaluated by the research team and the findings may be used for publication; however, any published or disseminated results will omit information that could potentially identify participants (name, date of birth, address and provincial health identifier number).